CLINICAL TRIAL: NCT06007079
Title: Clinical Data Collection Study Using CardioPulmonary Management System in Patients With Chronic Heart Failure
Brief Title: Clinical Data Collection Study Using CPM System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Analog Device, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ADI-NYP
Record Dates: First submitted 2023-08-18; First posted 2023-08-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device Use (Experimental): Patients will be given the CPM device to take home and use once daily
  Interventions: Device: CPM Device

INTERVENTIONS:
Device: CPM Device — Wearable monitor

SUMMARY:
This study will assess the deployment of the ADI CPM System in a home setting and determine the interoperability of the CPM System within existing care pathways for HF patients. Clinicians will be blinded to CPM generated data and acquired physiologic data will not be used in clinical decision-making. After conclusion of this phase, a retrospective review of CPM System-acquired data will be compared with changes in treatment and HF events. This retrospective review will inform the subsequent design of the interventional study that is planned. Study participation for each patient will last for six months inclusive of 5 months of daily CPM monitoring followed by 30 days of observation for HF-related events. The additional 30 days of medical record observation is intended to capture any events that might correspond to predictions made during the final weeks of CPM monitoring.

DETAILED DESCRIPTION:
The current investigation is designed to be an observational study of the feasibility of using the CPM system. Its goal is to familiarize the study team with the CPM system, uncover potential challenges in its deployment, assess its predictive ability, and ultimately define clinical protocols to react to CPM generated information. The next phase of investigation will be a pilot study of the efficacy of using the CPM system to prevent heart failure hospitalizations.

The patient will use the CPM device once daily during the first 5 months of the study. Patient records will be retrospectively reviewed over those 5 months plus an additional 30 days following the final CPM measurement to assess for any CHF-related events.

Baseline/Initial Visit (Visit 1):

At this visit, the start of the study, the information described in the "Baseline Assessments" section will be collected. The study will be re-described to the participant. The study team will then set up the device for the individual patient by making adjustments (as needed) to address patient specific anatomy, ensuring that the sensors are all contacting the appropriate chest areas, and confirming the measurements on the CPM Web application. The patient will be shown how to apply and replace the adhesive on the device, how to position the device, how to take a measurement with the device, and how to store the device on the Base Station. The trained provider will then register the baseline reading for the CPM device using the CPM Mobile App. Informational material about using the device, refreshing adhesives, and interpreting device LEDs and chimes will be provided to each patient. Each patient will be reminded to take a measurement with their CPM at the same time each day (preferably when they first wake up) and instructed to follow the medical regimen prescribed by their physician.

Between Visits:

Between visits, caregivers will not have any access to the data being collected on the CPM System. They should perform their usual standard of care on these patients. Participants will receive one call from the study team after 1 week of monitoring to check in about the progress of the study (i.e. if protocols are being followed correctly, if the CPM device is working properly, and if adherence is satisfactory). If the participant is found to have problems with the device, a follow up at week 2 can be scheduled. The check-in conversation topics should focus on any ease of use issues and address any technical barriers impacting compliance.

Follow-up Visit (Visit 2):

On this visit, which will take place at the end of the 5 months, the study team will make arrangements for the patient to return to the office for a check-up and return the device (the same tests as described in the "physical examination" section). Patients will also be asked about their perception on "ease of use", impact on day to day activities, and overall satisfaction with the CPM system. Thirty days following the last measurement the study team, will review the patients records for all HF related events and treatment changes. Study protocol will also include a phone call to the patient to inquire if they had any heart failure events during this time.

Post-Monitoring (Data review):

After the completion of the monitoring, the study team will analyze the de-identified data from the CPM system and correlate it with clinical events obtained from patients and their medical records. Threshold events flagged in the CPM data will then be compared to clinical data to determine the CPM's performance characteristics (sensitivity, specificity, PPV, NPV and AUC ROC), and median prediction time for HF events.

ELIGIBILITY:
Inclusion Criteria: Heart failure patients regardless of ejection fraction (HFpEF or HFrEF) with one or more of the following:

* NYHA Class III-IV
* NYHA Class II HF with one or more of the following:

  * Chronic Kidney Disease (eGFR<60)
  * HF hospitalization (defined as HF listed as the major reason for hospitalization) within 9 months prior to screening visit and NT-proBNP > 200 pg/ml for patients not in AF or > 600 pg/m for patients in AF on screening ECG
  * NT-proBNP > 300 pg/ml for patients not in AF or > 900 pg/ml for patients in AF on the screening visit ECG.
  * Chronic obstructive pulmonary disease (COPD)

Exclusion Criteria:

* Under 18 years of age
* Patients with severe COPD (GOLD stage III or IV)
* Chronic Kidney Disease (eGFR < 20)
* Limited mobility preventing application of device
* Cognitive impairments that would limit the application and proper use of the device
* Skin allergies or skin sensitivities to silicone-based adhesives
* Pregnancy
* Skin breakdown on the left chest or breast area
* Not willing to shave chest hair if needed to apply device
* Patients on chronic inotropic therapy
* Patients with any condition that might limit the survival to less than 1 year as assessed by the investigator
* No cellular coverage (Patient's Home)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Record number of heart failure events | 5 months
  A HF hospitalization is defined as any unplanned visit to a hospital, Emergency Department or Observation unit with a length of stay of at least 24 hours AND treatment with intravenous diuretics.
  Worsening heart failure is defined as having at least one sign or symptom of congestion including but not limited to: worsening dyspnea, orthopnea, PND, JVD, S3 gallop, pulmonary crackles, ascites or edema.
  Urgent treatment is defined as any use of intravenous diuretic therapy or an increased diuretic dosage (at least 2x baseline dose) and/or additional class of diuretics.
Sensitivity | 6 months
  Measuring the sensitivity of each parameter with respect to the ability to predict a CHF event. Sensitivity is defined as TP/(TP+FN) = True Positive/(True Positive+False Negative)
Specificity | 6 months
  Measuring the specificity of each parameter with respect to the ability to predict a CHF event. Specificity is defined as TN/(TN+FP) = True Negative/(True Negative+False Positive)

SECONDARY OUTCOMES:
Patient compliance | 5 months
  Percentage of days that patient completes a recording.
Data quality | 5 months
  Measuring valid data available (valid days of measurement / total number of measurements)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No